CLINICAL TRIAL: NCT00609479
Title: Comparison of External and Internal Fixationmethods for Distal Radius Fracture - a Randomized Study.
Brief Title: Comparison of Two Methods for Treatment of Colles´s Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: MD/PhD-stud. Jesper Ougaard Schønnemann, Orthopedic Research Unit, Regionhospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JOS-1; JOS-1
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Distal Radius Fracture; Colle´s Fracture
Keywords: Distal radius fracture; Colle´s fracture; Internal fixation; External fixation; DASH; PRWE
MeSH Terms: conditions — Wrist Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Internal fixation with Micronail. 41 patients.
  Interventions: Procedure: Osteosynthesis
- 2 (Experimental): External fixation with Hoffmann-II-non-bridging. 41 patients.
  Interventions: Procedure: Osteosynthesis

INTERVENTIONS:
Procedure: Osteosynthesis — 1. Micronail osteosynthesis. A cast for the first 14 days, thereafter starting physiotherapy. Control at weeks 1,2,5,12.
  2. Hoffmann-II-non-bridging osteosynthesis. Removal of device after 5 weeks. physiotherapy starts at 14 days. Control at weeks 1,2,5,12.

SUMMARY:
The purpose of this study is to compare two different fixationmethods for fractures of the wrist(distal radius fractures). We are comparing an external fixation (Hoffmann-II-non-bridging) vs. an internal fixation(Micronail). Primary endpoint is patient satisfaction as scored by the DASH-questionnaire.Secondary followup is X-rays, strength, PRWE-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Fracture Older type 2.
* Fracture Older type 3.

Exclusion Criteria:

* Fractures older than 3 weeks.
* Pregnancy.
* Seq. after previous fracture.
* Distal fragments volar cortex < 10 mm.
* Open fracture larger than Gustillo 1.
* Disability due to other illness.
* Congenital abnormity or injury/disease in the affected extremity.
* Not capable of mentally/physically to cooperate.
* Not able to go to followup on the operating hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
DASH-questionnaire | 3 months

SECONDARY OUTCOMES:
PRWE-questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD; PhD; Prof., Study Chair — Department of Orthopedics, University of Aarhus, Denmark
Locations (3):
- Denmark (3):
  - Regionhospital Herning, Herning
  - Regionhospital Holstebro, Holstebro
  - Regionhospital Viborg, Viborg